CLINICAL TRIAL: NCT00047788
Title: A Phase Two Study of ZD6474 in Patients With Relapsed Multiple Myeloma
Brief Title: Efficacy Study of ZD6474 to Treat Multiple Myeloma Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6474IL/0004; IND.145(Canada); NCT00052741 (obsolete NCT alias)
Record Dates: First submitted 2002-10-18; First posted 2002-10-21 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — vandetanib

INTERVENTIONS:
Drug: ZD6474
Drug: VEGF-receptor tyrosine kinase (KDR)

SUMMARY:
The primary objective is to assess the efficacy of ZD6474 when given orally to patients with relapsed multiple myeloma. A minimum of 15 and a maximum of 30 evaluable patients will be entered on study

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma.
* Patients must have a minimum serum M-protein level >=10g/L on serum protein electrophoresis or for patients with light chain only disease, a minimum Bence-Jones protein of 1g/24 hr.
* Patients must have received prior treatment for multiple myeloma: patients may have received 1 or 2 prior regimens of oral alkylating based chemotherapy and must have relapsed following treatment (>= 3 months) OR patients may have relapsed following high dose chemotherapy and SCT as first line treatment provided they have not had any other treatment.
* Lab at inclusion of AGC >= 1.0 x10_9/L and platelets >= 50 x10_9/L Bilirubin, AST and/or ALT <= 1.5 x UNL; creatinine < 2 x UNL, Potassium >= 4.0 mmol/L; calcium and magnesium within normal limits·
* Patients may not have had > 2 prior regimens of chemotherapy and/or prior thalidomide treatment.
* Patients may not have had any non-alkylating based chemotherapy.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for >= 5 years.
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test within 7 days prior to registration and must be using effective contraception throughout the study.
* Patients who have relapsed during treatment with oral alkylating chemotherapy.
* Patients who have received more than 2 prior regimens of chemotherapy.
* Patients who have received excluded medication or have excluded medical conditions.
* Patients who have received any non-alkylating based chemotherapy regimens as initial therapy, or as therapy for recurrent disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-10; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Research Site, New York, New York, United States
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec